CLINICAL TRIAL: NCT06621706
Title: Ultrasound Assessment of Gastric Volume in Diabetic Versus Non-Diabetic Term Pregnant Women Undergoing Elective Cesarean Section: A Prospective Randomized Clinical Trial
Brief Title: Ultrasound Assessment of Gastric Volume in Diabetic Versus Non-Diabetic Term Pregnant Women Undergoing Cesarean Section
Status: Recruiting | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Dina Mahmoud Fakhry, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Management, Beni-Suef University
Other Study IDs: FMBSUREC/01092024/Fakhry
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Aspiration; Gastric Content Aspiration
Keywords: Diabetic; Gastric ultrasonography; Pregnant
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic term pregnant group: Compare the antral cross-sectional area (CSA) with gastric ultrasonography and estimated gastric volumes
  Interventions: Device: Gastric ultrasonography
- Non-diabetic term pregnant group: Compare the antral cross-sectional area (CSA) with gastric ultrasonography and estimated gastric volumes
  Interventions: Device: Gastric ultrasonography

INTERVENTIONS:
Device: Gastric ultrasonography — Women will be requested to fast 2 hours for clear drinks, 6 hours for a light meal, and 8 hours for a meal high in fried or fatty content prior to their next antenatal clinic visit.
  On the day of assessment, fasting and dietary compliance will be confirmed individually with each woman and Gastric ultrasonography will be performed after sex and eight hours of fasting food.
  Women will be first scanned in a semi-recumbent (45 degrees head up) supine position, followed by a semi-recumbent (45 degrees head up) right lateral position (RLP). In both positions the gastric antrum will be identified in the sagittal plane with its internal anatomical landmarks identified, i.e. the left lobe of the liver anteriorly and the abdominal aorta posteriorly.

SUMMARY:
The aim of the work to compare estimated gastric volumes through ultrasound in fasting diabetic and non-diabetic pregnant women scheduled for caesarean section.

DETAILED DESCRIPTION:
Fasting is a mandatory requirement prior to elective anesthesia and is intended to reduce gastric fluid volume and the risk of aspiration of gastric contents and subsequent organ injury. Aspiration of gastric contents during perioperative period is a grave complication with significant morbidity and mortality and its severity depends upon the gastric volume and nature of the aspirate.

A high-risk stomach refers to a gastric volume associated with an increased risk of pulmonary aspiration and is defined in most published literature as the presence of any solid or liquid content >1.5 mL/kg Pregnant women have been considered to be at particular risk of aspiration syndromes as a consequence of physiological changes during pregnancy which lead to relaxation of lower oesophageal sphincter and mechanical upward displacement of the stomach by the enlarged uterus.

European Society of Anaesthesiology (ESA) recommends fasting for ≥2 hours after clear liquids and 6 hours after light meals before elective surgery, including in pregnant patients. In contrast, the American Society of Anesthesiology guidelines specifically exclude pregnant women and the Society for Obstetric Anesthesia and Perinatology taskforce recommended a fasting period of 6-8 hours, depending on the nature of food ingested.

Diabetic patients can present with diabetic gastropathy, an autonomic neuropathy associated with delayed gastric emptying in the absence of gastric outlet obstruction tend, predisposing them to increased risk of aspiration as compared to non-diabetic patients.

To date, standard fasting guidelines for people with diabetes are still up for debate.. European Society of Anaesthesiology (ESA) 2011 Fasting guidelines state that diabetic patients can follow the same guidelines as healthy adults, While American Society of Anesthesiologists (ASA) in 2017 fasting guidelines mentioned that the standard eight hours fasting may not apply or may need to be modified for patients with coexisting diseases or conditions that can affect gastric emptying or fluid volume.

With the advent of portable ultrasound machines, performing point-of-care ultrasound has become relatively easy and feasible. Gastric ultrasound examination is finding a place as a point-of-care tool for aspiration risk assessment. It can identify the nature and the volume of the gastric content, i.e., empty, clear fluid and solid and when clear fluid is present, its volume can be quantified.

In this study, we will analyse the stomach contents of Non-labouring term pregnant women after six and eight hours of fasting, using previously described qualitative and quantitative ultrasonographic assessments.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women undergoing elective caesarean section
* aged between 18-40 years
* belonging to ASA II-III
* gestational age greater than 37 weeks
* BMI< 35 kg/m2

Exclusion Criteria:

* patients who refuse to give consent
* patients taken to surgery on an emergency basis, -pregnant patients with upper gastrointestinal (GI) diseases and pathologies
* patients with a history of using medications that affect gastrointestinal motility (e.g., opioids), severe organ dysfunction
* pre-existing neurological deficits, intellectual disabilities and anatomical deformities.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Eligible 140 patients are aged from 18-40 years, with an American Society of Anaesthesiologists (ASA) physical status of II-III, and are scheduled to undergo elective caesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
mean antral cross-sectional area of stomach | 8 hours of fasting
  mean antral cross-sectional area of stomach after 8 h of fasting in term pregnant diabetic and non-diabetic women undergoing elective caesarean section.

SECONDARY OUTCOMES:
the mean antral cross-sectional area of stomach | 6 hours of fasting
  mean antral cross-sectional area of stomach after 6 h of fasting presence of solid food contents in the gastric antrum,
gastric antral grade | 6 and 8 hours of fasting
  The qualitative assessment of the gastric contents will be also done for presence of any clear fluid or solid food particles and a gastric antral grade, as described by Perlas et al. was designated based on the presence of fluid as follows: Grade 0 = absence of fluid in both supine and RLP; Grade 1 = fluid in RLP only; Grade 2 = fluid in both supine and RLPs

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Fakhry, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University hospital, Banī Suwayf, Beni Suweif Governorate, Egypt